CLINICAL TRIAL: NCT04938778
Title: Prolonged Nightly Fasting (PNF) in Older Adults With Age-related Cognitive Decline: A Pilot Study Exploring Changes in Neurocognitive Function (Public Name:Think FAST)
Brief Title: Think FAST Research Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Darith James, Postdoctoral Researcher, Arizona State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00012888
Record Dates: First submitted 2021-03-10; First posted 2021-06-24 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Age-related Cognitive Decline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): 8 week 14 hour prolonged nightly fasting intervention.
  Interventions: Other: PNF

INTERVENTIONS:
Other: PNF — PNF Participants will engage in 8 weeks of 14 hours per night fasting

SUMMARY:
To test a 14-hour prolonged nightly fasting (PNF) protocol in a group of older adults (≥ 65 years old) with self-identified age-related cognitive decline (ARCD) on the primary outcome of neurocognitive function and performance as measured by objective outcomes. The investigators will use an 8-week single group pre-post pilot study design to measure outcomes related to neurocognitive function and performance and cardiometabolic risk factors (i.e., sleep disturbances, body mass index).

ELIGIBILITY:
Inclusion Criteria:

* 65 or older
* Self-identified age-related cognitive decline (ARCD)
* Has a text capable phone and access to wifi

Exclusion Criteria:

* Diagnosed with an eating disorder in the past 20 years
* Works a night shift
* Cannot participate in a 14 hour fast
* Has diabetes

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Memory and Attention Phone Screener (MAPS) | 8 weeks
  Cognitive Function and Performance Test.

SECONDARY OUTCOMES:
Rapid Eating Assessment for Participants Scale (REAPS) | 8 weeks
  Scale to asses eating behaviors. The scale has a minimum of 13 and a maximum of 39. Higher scores indicate higher diet quality.
Insomnia Severity Index (ISI) | 8 weeks
  Scale to asses insomnia symptoms. The scale has a minimum of zero and maximum of 28 where zero would be absence of insomnia and 28 would be severe insomnia.
Mindful Eating Scale (MES) | 8 weeks
  Scale to asses behaviors related to mindful eating. Each item has a minimum of zero and a maximum of 4 where 4 means less eating awareness.
Creature of Habit Scale (COHS) | 8 weeks
  Scale to asses routine habits. Each item has a minimum of zero and a maximum of 4 where 4 means a more habitual nature.
Salivary Cortisol | 8 weeks
  Measure of cortisol via participant saliva samples.
Body Mass Index (BMI) | 8 weeks
  Self-reported body measurements .

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States